CLINICAL TRIAL: NCT01164514
Title: A Randomized, Partial-Blinded, Placebo-Controlled, Phase I Safety and Immunogenicity Study in Healthy Subjects of Detoxified J5 Core Glycolipid/ Group B Meningococcal Outer Membrane Protein Vaccine for Gram Negative Bacterial Sepsis Administered With and Without Synthetic CPG Oligodeoxynucleotide 7909 Adjuvant
Brief Title: Detoxified J5 Core Glycolipid/ Group B Meningococcal Outer Membrane Protein Vaccine for Gram-negative Bacterial Sepsis Administered With and Without Synthetic CPG Oligodeoxynucleotide 7909 Adjuvant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-086; N01AI80057C
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2012-08

CONDITIONS: Bacterial Sepsis
Keywords: bacterial sepsis, septicemia, vaccine
MeSH Terms: conditions — Sepsis | interventions — ProMune

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group 1 - vaccine alone (Active Comparator): 8 subjects to receive vaccine (10 mcg) alone on Days 0, 29 and 59.
  Interventions: Biological: J5-OMP Vaccine
- Group 3 - vaccine + CPG 7909 (250 mcg) (Experimental): 8 subjects to receive vaccine (10 mcg) with 250 mcg of adjuvant on Days 0, 29 and 59.
  Interventions: Biological: CPG 7909; Biological: J5-OMP Vaccine
- Group 2 - vaccine + CPG 7909 (500 mcg) (Experimental): 8 subjects to receive vaccine (10 mcg) with 500 mcg of adjuvant on Days 0, 29 and 59.
  Interventions: Biological: CPG 7909; Biological: J5-OMP Vaccine
- Group 4 - Placebo (Placebo Comparator): 4 subjects to receive normal saline (placebo) on Days 0, 29 and 59.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CPG 7909 — CPG 7909 is a synthetic oligodeoxynucleotide used as an adjuvant and administered at 2 different dosages: 250 mcg and 500 mcg.
  Arms: Group 2 - vaccine + CPG 7909 (500 mcg); Group 3 - vaccine + CPG 7909 (250 mcg)
Biological: J5-OMP Vaccine — J5-OMP vaccine 10 mcg to be administered with and without CpG 7909 adjuvant 250 or 500 mcg, intramuscularly on Days 0, 29 and 59.
  Arms: Group 1 - vaccine alone; Group 2 - vaccine + CPG 7909 (500 mcg); Group 3 - vaccine + CPG 7909 (250 mcg)
Drug: Placebo — Normal saline.
  Arms: Group 4 - Placebo

SUMMARY:
The purpose of this study is to test the safety of an experimental vaccine against sepsis (infection of the blood) alone and with an experimental adjuvant (a substance that may improve vaccine effectiveness). This study will also find out how well antibodies are made after receiving vaccine alone or vaccine combined with adjuvant. Participants will include up to 34 healthy volunteers between the ages 18-50 years. Participants will be randomly assigned to 1 of 4 groups to receive vaccine alone, vaccine with adjuvant (2 different dosages) or placebo (inactive substance). Participants will receive 3 vaccinations at different times during the study (Day 0, Day 29 and Day 59). Study procedures will include blood samples, urine samples, electrocardiogram (measures heart activity) and a completion of a memory aid to document side effects. Participation will involve 16 clinic visits and 3 follow-up telephone calls over 12 months.

DETAILED DESCRIPTION:
Invasive Gram negative bacterial infection resulting in sepsis continues to command substantial morbidity and mortality despite effective antibiotics and modern intensive care. It has been estimated that there are 300,000 cases per year in the United States. The emergence of multiple antibiotic resistant strains of bacteria adds to the urgency of finding novel therapies for the treatment of gram negative sepsis. Sepsis is a systemic inflammatory condition characterized by fever, hypotension, tachypnea, and tachycardia which can lead to multiple organ/system failure and ultimately death. This study is a randomized, partial blinded, placebo-controlled phase I safety and immunogenicity study in healthy subjects of detoxified J5 core glycolipid/ group B meningococcal outer membrane protein vaccine for gram-negative bacterial sepsis administered with and without synthetic unmethylated cytosine-guanosine motif (CPG) oligodeoxynucleotide 7909 adjuvant. The primary objective of this study is to establish the safety and tolerability of the combination of vaccine and CPG 7909. The secondary objective of this study is to determine if the combination of vaccine with the CPG 7909 is more immunogenic than vaccine alone. One dosage level of vaccine based on lipopolysaccharide (LPS) content will be studied in a three-dose regimen administered intramuscularly (IM). Since prior experience indicates no significant differences in immunogenicity response between the 10 and 25 microgram (mcg) doses of vaccine, researchers will test the 10 mcg dose. Researchers will also use 2 different doses of the CPG 7909 adjuvant (500 mcg and 250 mcg). There will be a control group that receives normal saline (NS) alone (placebo). The purpose of this study is to assess whether or not this vaccine is safe and well tolerated when given with an adjuvant, CPG 7909. The other goal of this study is to ascertain whether or not the combination of vaccine and adjuvant induces a more robust antibody response to the vaccine than is observed with the vaccine alone. The study population will include approximately 28-34 healthy subjects ages 18-50 years, inclusive, recruited from existing pool of Center for Vaccine Development (CVD) subjects. Subjects will be randomized to one of four study groups: (Group 1) 10 mcg vaccine alone; (Group 2) 10 mcg vaccine plus 500 mcg CPG 7909; (Group 3) 10 mcg vaccine plus 250 mcg CPG 7909; and (Group 4) placebo (normal saline). After blood is obtained for pre-vaccination antibody levels, subjects will receive 3 vaccinations at Day 0, 29 and 59. Subjects will be followed for safety (both clinical signs and symptoms and laboratory tests) and antibody response (anti-core glycolipid antibody by enzyme linked immunosorbent assay [ELISA], and opsonophagocytic response). Assessments for reactogenicity will be done for 60 minutes post vaccination and on the first and second days after each vaccination at the CVD and via 8 day memory aid, to be completed by the subject, after each vaccination. An electrocardiogram (EKG) will be performed after each vaccination. Blood sampling will be performed on Days 0, 14, 36, 66, 120, 180, and 365 to measure the immunogenicity of the vaccine with and without adjuvant and for antibody screening. A safety evaluation will be done by telephone on Day 90, Day 150 and Day 239, and a final safety antibody and immunogenicity evaluation will be done during the clinic visit at Day 365.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18-50 years, inclusive.
* The subject has provided written informed consent prior to any study procedures.
* Able to attend scheduled visits and comply with trial procedures.
* The subject is in good health as determined by vital signs [heart rate <100 beats per minutes (bpm); blood pressure: systolic greater than or equal to 90 mm Hg and less than or equal to 140 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature <100.0 degrees Fahrenheit], medical history to ensure stable medical condition and a physical examination based on medical history. A stable medical condition is defined as no recent change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company, etc, or is done for financial reasons, as long as in the same class of medication, will not be considered a violation of the inclusion criterion. Any change to prescription medication due to improvement of a disease outcome will not be considered a violation of the inclusion criterion.
* Women of child-bearing potential or their partners must be surgically sterile or must agree to use an effective method of contraception and agree to remain on that same method through Day 120. Male subjects or their partners must be surgically sterile or must agree to use effective contraception through Day 120. (e.g. hormonal contraceptives initiated at least 30 days prior to receipt of vaccine, intrauterine devices (IUDs), diaphragm in combination with contraceptive jelly, condoms in combination with contraceptive jelly, cream, or foam; or vasectomized partner).
* Have normal laboratory values for hemoglobin, white blood cells (WBC) and platelets, absolute neutrophil count (ANC), absolute lymphocyte count (ALC) obtained from the complete blood count (CBC), and serum glucose and thyroid stimulating hormone (TSH). Serum alkaline phosphatase, aspartate aminotransferase (AST), alanine transferase (ALT), blood urea nitrogen (BUN), C-reactive protein (CRP) and creatinine are not to exceed the upper limit of normal, and urinalysis must be normal on day of screening visit.
* Must have a negative pregnancy test at screening (serum) and negative pregnancy test (urine) on days of vaccination, with known results prior to vaccination.
* Subject agrees to avoid non-study related blood donation for 1 year following the last immunization.

Exclusion Criteria:

* History of allergy or severe reaction to any vaccine or vaccine components or unmethylated cytosine-guanosine motif (CPG) components.
* Acute illness or fever >/= 38 degrees Celsius/100.4 degrees Fahrenheit within a week prior to each vaccination.
* Prior receipt of any Group B meningococcal outer membrane protein (OMP) vaccine.
* Previous receipt of oligodeoxynucleotide adjuvant including CPG.7909.
* Immunosuppression as a result of underlying illness or treatment.
* Use of oral steroids, parenteral steroid or high-dose inhaled (>800 mcg/day of beclomethasone dipropionate or equivalent) within 30 days prior to each vaccination.
* Acute or chronic condition that (in the opinion of the investigator) would render vaccination unsafe or would interfere with the evaluation of responses including, but not limited to the following: cardiovascular, known chronic liver disease, significant renal disease, chronic lung diseases, unstable neurologic disorder.
* Receipt of immunoglobulin or other blood product within 3 months prior to enrollment.
* Current excessive use of alcohol or drug dependence (>8 ounces of liquor or >96 ounces of beer/day) or a history of alcohol or drug abuse in the 5 years prior to enrollment.
* History of meningococcal infection.
* Diagnosed autoimmune condition in either subject or immediate family member.
* Under the care of a physician for a diagnosed psychiatric condition.
* Women who are pregnant or breast feeding.
* Women with a current or recent (i.e. within two half-lives) history of diuretic or promethazine use.
* The subject is immunosuppressed as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* The subject has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematologic malignancy. An active neoplastic disease is defined as treatment for neoplastic disease within the past 5 years.
* The subject has received an inactivated vaccine within the 2 weeks or a live vaccine within the 4 weeks prior to enrollment in this study or plans to receive another vaccine in the next 28 days.
* The subject is currently participating in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study.
* The subject has a current or life-time diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis.
* The subject has been hospitalized within the past 2 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* The subject is receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug, are not diagnosed with depression and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* The subject has a known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* The subject has an electrocardiogram (EKG) showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any nonsinus rhythm excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
* The subject has a history of working in an infectious disease laboratory.
* Any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render them unable to comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Clinical measures: severity and duration of systemic and local adverse events (AEs), and vaccine-related serious adverse events (SAEs) | Solicited local and systemic adverse events (AEs) within 8 days post vaccination (Day 0-7); vaccine-related serious adverse events (SAEs) throughout the course of the study.

SECONDARY OUTCOMES:
Immunogenicity measures: mean fold-increase in anti-J5 detoxified lipopolysaccharide (dLPS) IgG and IgM levels in serum and percent of subjects having >/= 4-fold IgG and IgM antibody titer response, time to seroconversion. | Blood sampling Days 0, 14, 36, 66, 120, 180 and 365.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical System - General Clinical Research Center (GCRC), Baltimore, Maryland, United States

REFERENCES:
- [Derived] Cross AS, Greenberg N, Billington M, Zhang L, DeFilippi C, May RC, Bajwa KK. Phase 1 testing of detoxified LPS/group B meningococcal outer membrane protein vaccine with and without synthetic CPG 7909 adjuvant for the prevention and treatment of sepsis. Vaccine. 2015 Nov 27;33(48):6719-26. doi: 10.1016/j.vaccine.2015.10.072. Epub 2015 Oct 26. PMID 26514420